CLINICAL TRIAL: NCT00591292
Title: IBL1002:Phase I Study of Indibulin in Advanced Solid Tumors
Brief Title: Phase I Study in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL1002
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
Keywords: cancer; tumor; solid tumor; advanced tumor
MeSH Terms: conditions — Neoplasms | interventions — indibulin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: indibulin

INTERVENTIONS:
Drug: indibulin — Dose escalation of indibulin given twice daily for up to 6 months
  Other Names: ZIO-301

SUMMARY:
Dose escalating study of orally administered indibulin at twice daily schedule in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria

1. Subjects with histological or cytological confirmation of advanced cancer, refractory to standard therapies for their condition
2. ≥ 18 years of age
3. ECOG performance score ≤ 2 (see Appendix 3)
4. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines (See Appendix 4). If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions MUST not have been in a previously irradiated field or injected with biological agents.
5. Life-expectancy ≥ 12 weeks
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted < 2 weeks prior to Baseline:

   * Creatinine ≤ 1.5 X upper limit of normal (ULN) OR a calculated creatinine clearance ≥ 50 cc/min
   * Total bilirubin ≤ 1.5 X ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 X ULN
   * White blood cell count ≥3.0 x 109/L
   * Absolute Neutrophil Count (ANC) ≥1.5 x 109/L
   * Platelets ≥100 x 109/L
   * Hemoglobin ≥ 10 g/dL
7. Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee with jurisdiction over the site.

Exclusion Criteria

1. New York Heart Association (NYHA) functional class ≥3 or myocardial infarction within 6 months (see Appendix 5)
2. Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation
3. Pregnant and/or lactating female (a reliable method of contraception must be used in all men and in women of childbearing potential during the study and for 3 months after last study drug administration).
4. Uncontrolled systemic infection (documented with microbiological studies)
5. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry. Mitomycin C or nitrosureas should not be given within 6 weeks of study entry.
6. Radiotherapy during the study or within 3 weeks of study entry
7. Surgery within 4 weeks of start of study drug excluding tumor biopsy for pharmacodynamic parameters
8. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
9. History of an invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer
10. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
11. Any condition that is unstable or which could jeopardize the safety of the subject and his/her compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, Study Director — Alaunos Therapeutics
Locations (1):
- Santa Monica, California, United States

REFERENCES:
- [Derived] Kapoor S, Srivastava S, Panda D. Indibulin dampens microtubule dynamics and produces synergistic antiproliferative effect with vinblastine in MCF-7 cells: Implications in cancer chemotherapy. Sci Rep. 2018 Aug 17;8(1):12363. doi: 10.1038/s41598-018-30376-y. PMID 30120268